CLINICAL TRIAL: NCT01875263
Title: Efficacy of a Short-term Sequential Therapy Versus Intravenous Standard Treatment for Patients With Non-complicated Catheter Related Bacteremia by Methicillin- Susceptible S.Aureus.
Brief Title: Efficacy of a Short-term Sequential Therapy in Non-complicated Catheter Related Bacteremia by Methicillin- Susceptible S.Aureus.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Not participants inclusion
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPS-COL-2013-06; 2013-000511-24 (EudraCT Number)
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Staphylococcus
Keywords: catheter-related bacteremia, SAMS; catheter related bacteremia; susceptible; aureus meticillin
MeSH Terms: conditions — Short Stature, Auditory Canal Atresia, Mandibular Hypoplasia, Skeletal Abnormalities; Disease Susceptibility | interventions — Cloxacillin; Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Cloxacillin 2g / 4 hours iv, 5 days followed levofloxacin 500 mg po / 24, 9 days.
  Interventions: Drug: Cloxacilin; Drug: Levofloxacin
- Control (Active Comparator): Cloxacillin 2g / 4 hrs iv 14 days
  Interventions: Drug: Cloxacillin

INTERVENTIONS:
Drug: Cloxacilin — 2g/4 hours i.v., 5 days
  Arms: Experimental
Drug: Cloxacillin — 2g/4h 14 days Standard therapy
  Arms: Control
Drug: Levofloxacin — 500 mg v.o./24h, 9 days
  Arms: Experimental

SUMMARY:
Evaluate the efficacy of a sequential regimen of 14 days in patients with catheter-related bacteremia by S. aureus methicillin-susceptible, selected based on a pre-established clinical and microbiological criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years with a minimum weight of 40 kg.
* Microbiological Isolation of S. aureus susceptible to meticillin.
* Start antibiotic treatment with drugs active against S. aureus within 72 hours from the onset of clinical manifestations.
* Women of childbearing potential, negative pregnancy test negative serum or urine or statement is not pregnant.
* Prescription prior treatment must be independent and decoupled patient inclusion in the study, corresponding exclusively to clinical practice.

Exclusion Criteria:

* Polymicrobial bacteremia.
* Neutropenic patients.
* Patients addicted to intravenous drugs.
* Patients with malignancies with expected survival less than 6 months.
* Severe allergy to beta-lactams or fluoroquinolones.
* Creatinine clearance <20ml/min.
* Need for hemodialysis, peritoneal dialysis or plasmapheresis.
* Clinical signs of deep infection in the first five days of treatment (mucocutaneous lesions suggestive of IE, embolic events, suppurative thrombophlebitis.
* Predictors of bacteremia complicated:
* Positive blood cultures for 48-96 hours of starting treatment antistaphylococcal
* Clinical Instability
* Signs of sepsis or persistent fever at day 4 of treatment
* Existence of valvular or vascular prosthetic joints, vascular catheter not removed within three days
* Heart disease predisposing to endocarditis.
* Patients presenting diagnosis concomitant infection by another organism.
* Pregnant or breast-feeding.
* Patients with epilepsy.
* Patients with a history of tendon disorders related to fluoroquinolone administration.
* Not have signed informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Reduce the rate of late complications of catheter-related bacteremia by S. aureus methicillin sensitive below 2%. | 18 months

SECONDARY OUTCOMES:
Reducing hospital stay associated with the treatment of uncomplicated bacteremia MS S. aureus. | 18 months
Reduce the transesophagic echocardiography | 18 months
  Increase efficiency in the management of patients with bacteremia due to MS S. aureus, reducing the number of echocardiographic evidence

CONTACTS AND LOCATIONS:
Locations (11):
- Spain (11):
  - Hospital de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Complejo Hospitalario de Huelva, Huelva
  - Hospital Can Misses, Ibiza Town
  - Hospital Comarcal Carlos Haya, Málaga
  - Hospital de Antequera, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitario Virgen del Rocío, Seville